CLINICAL TRIAL: NCT00573560
Title: A Feasibility Trial to Evaluate the VPD Implant System - Percutaneous Ventricular Restoration in Chronic Heart Failure Due to Ischemic Heart Disease
Brief Title: Safety Study of the Ventricular Partitioning Device (VPD) Implant System in Heart Failure Patients
Acronym: PARACHUTE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CardioKinetix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US PARACHUTE Protocol
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2014-07

CONDITIONS: Heart Failure
Keywords: Heart failure; percutaneous; interventional cardiology; apical remodeling; LV dilatation; akinesis; dyskinesis
MeSH Terms: conditions — Heart Failure; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: VPD Implant System — Percutaneous introduction using standard catheterization techniques of the VPD Implant.

SUMMARY:
The CardioKinetix Ventricular Partitioning Device (VPD) is intended to isolate the malfunctioning portion of the left ventricle in patients with symptoms of heart failure due to ischemic heart disease. By isolating the malfunctioning portion of the left ventricle, it is hypothesized that the left ventricle will pump more effectively.

ELIGIBILITY:
Inclusion Criteria:

1. Akinesis or dyskinesis due to myocardial infarction limited to anteroapical region
2. Diagnosis of heart failure for a minimum of 6 months prior to enrollment
3. NYHA Class at time of enrollment, either:

   * NYHA Class III or IV - if predominant during the 3-month period prior to enrollment
   * NYHA Class II - if diagnosed with NYHA Class III or IV during 3-month period prior to enrollment and ≥ 1 hospitalization for heart failure during 12-month period prior to enrollment
4. LVEF ≤ 40% as measured by echocardiography
5. Left ventricle must have appropriate anatomy as measured by Cardiac CT per the VPD Implant sizing criteria described in the device's Instructions For Use
6. Eligible for cardiac surgery
7. Between 18 and 74 years of age (inclusive)
8. Receiving appropriate medical treatment for heart failure according to the ACC/AHA 2005 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult during the three months prior to enrollment
9. Female patients with childbearing potential must have a negative pregnancy test (within 7 days of the procedure) and must agree not to attempt to become pregnant during the course of the study
10. Provide written informed consent
11. Agree to the protocol-required follow-up

Exclusion Criteria:

1. Myocardial ischemia requiring PCI or CABG
2. Acute MI (see MI definition) within 60 days of enrollment or patients with suspected evolving MI at time of enrollment
3. Cardiogenic shock within 72 hours of enrollment
4. Revascularization procedure (PCI or CABG) within 60 days of enrollment
5. Patient has received a CRT device within 60 days of enrollment
6. Patient diagnosed with significant valve disease (AI >1+; MR >2+) which may or may not require surgery
7. Patient has received an ICD within 60 days of enrollment
8. Patient has received a pacemaker within 60 days of enrollment
9. History of aborted sudden cardiac death, if patient has not received an ICD and has potentially lethal ventricular arrhythmia, VT or VF
10. Patients with a history or a current diagnosis of either persistent or paroxysmal atrial fibrillation as well as patients who present with a contraindication to oral anticoagulant therapy
11. Aortic valve replacement or repair
12. Resting systolic blood pressure is more than 180 mmHg or less than 90 mmHg
13. Resting heart rate more than 120 bpm
14. Cardiac CT or echocardiographic evidence of thrombus in the left ventricle or left atrium
15. History of bleeding diathesis or a major coagulopathy (i.e. platelet count < 100,000 plts/ml whole blood; PTT or PT > 1.3 times control value)
16. GI bleed requiring transfusion within the past 3 months
17. Patient has suffered a stroke within the past 6 months
18. Evidence of severe calcification in the VPD Implant attachment zone
19. Evidence of a significant sub-aortic obstruction ("left moderator band") in the area of implant
20. History of Kawasaki's disease
21. Patient has received a heart, lung, liver and/or kidney transplant
22. Patient on dialysis or expected to require hemodialysis within 12 months
23. Patient has chronic liver disease
24. Patient has received intracardiac gene therapy or stem cell therapy
25. Creatinine > 2.5mg/dl or impaired renal function that places patient at risk of contrast induced renal failure
26. Hypersensitivity to contrast media
27. Allergy or contraindication to clopidogrel or aspirin
28. Evidence of ongoing infection (fever with temperature > 38°C and/or WBC > 15,000)
29. Co-morbidities associated with a life expectancy of less than 12-months or there are factors making echo and clinical follow-up difficult (no permanent address, etc.)
30. Patient is currently participating in another investigational device or drug research study for which the follow-up period is not complete

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Assessment of safety defined as the successful delivery and deployment of the VPD Implant through 6 month follow up without the occurrence of Major Adverse Cardiac Events (MACE) related to the investigational device. | 6 months

SECONDARY OUTCOMES:
Preliminary Effectiveness Measurements at 6 months - Change in LV volume indices (LVESVI, LVEDVI, EF) - Change in 6 minute walk and VO2 max - Cardiovascular mortality and morbidity inclusive of hospitalization for HF, MI and stroke | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: William T Abraham, MD, Principal Investigator — Ohio State University
Locations (7):
- United States (6):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Northwestern University Medical Center, Chicago, Illinois
  - Mission Hospitals, Asheville, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Texas Heart Institute, Houston, Texas
- Dedinje Cardiovascular Institute, Belgrade, Serbia

REFERENCES:
- [Derived] Costa MA, Mazzaferri EL Jr, Sievert H, Abraham WT. Percutaneous ventricular restoration using the parachute device in patients with ischemic heart failure: three-year outcomes of the PARACHUTE first-in-human study. Circ Heart Fail. 2014 Sep;7(5):752-8. doi: 10.1161/CIRCHEARTFAILURE.114.001127. Epub 2014 Jul 18. PMID 25037310